CLINICAL TRIAL: NCT06623201
Title: Blue-Light Photodynamic Therapy and Sonidegib for Multiple Basal Cell Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nathalie Zeitouni (Other)
Responsible Party: Sponsor-Investigator, Nathalie Zeitouni, Sponsor-Investigator, US Dermatology Partners, Phoenix
Organization: US Dermatology Partners, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT-MDS-BCC-24
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Basal Cell Carcinoma (BCC)
Keywords: Basal cell carcinoma; Levulan; PDT
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Open-label study where all participants receive the same treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Blue-Light Photodynamic Therapy and Sonidegib (Experimental): All subjects will receive Sonidegib (ODOMZO) 200mg by mouth every day on an empty stomach (1 hour before or 2 hours after a meal) for 3 months, and PDT with topical application of ALA for a total of 3 sessions. PDT will be first administered at Visit 3 (Day 7), Visit 4 (Day 45), and Visit 5 (Day 75).
  Interventions: Drug: aminolevulinic acid HCL (ALA); Device: BLU-U device model 4170E

INTERVENTIONS:
Drug: aminolevulinic acid HCL (ALA) — Prior to ALA application, the areas will be cleaned with alcohol and debrided gently with prep tape. ALA will then be applied to each of the study lesions and allowed to incubate for 3 hours with occlusion prior to the PDT.
Device: BLU-U device model 4170E — Participants will be subjected to dose illumination with blue light (BLU-U Model 4170E) at a power fluence of 20 mW/cm2 for a total time of 16 minutes and 40 seconds (1,000 seconds). This will result in a total light delivery dose of 20 J/cm2.

SUMMARY:
This research study is testing combination Blue-light photodynamic therapy and Sonidegib as a possible treatment for people with multiple basal cell carcinoma lesions.

Basal cell carcinoma lesions are typically treated by freezing the lesion or surgically removing the lesion. These types of treatment can cause scarring. Photodynamic therapy uses light along with a drug applied to the skin to kill the cancer cells and cause them to break apart. The light used can cause the skin to feel warm, but does not cause scarring.

DETAILED DESCRIPTION:
Blue light PDT has shown some success in treating BCCs, but more research is needed to evaluate this treatment modality further. The objective of this study is to evaluate the safety and efficacy of using photodynamic Therapy with Sonidegib for the treatment of multiple nodular basal cell carcinomas. Participants who meet eligibility criteria at baseline will receive Sonidegib 200 mg by mouth every day for 3 months. Participants will undergo three PDT sessions with topical application of ALA at Day 7, Day 45, and Day 75.

The drug applied to the skin before the light treatment is an FDA approved drug called Levulan and has no known side effects. The light used to treat the lesion is blue light illumination using the BLU-U Blue Light Photodynamic Therapy Illuminator (Levulan-PDT). This treatment regimen is approved by the FDA to treat actinic keratoses, but is not approved to treat basal cell carcinoma. Use of the light can feel warm and may sting.

Sonidegib (Odomzo) is a compound that was approved by the US Food and Drug Administration in July 2015 as a treatment option for BCC. Patients on Sonidegib may experience leg cramps, taste disturbance, or alopecia

ELIGIBILITY:
Patients will be included in the study based on the following criteria:

1. Male or females, at least 18 years of age.
2. Diagnosis of BCC with at least 3 nodular lesions that measure 0.5 cm to 5 cm in diameter, located on the head and neck, trunk or extremities.
3. Diagnosis must be confirmed clinically at baseline with 1-3 lesions having been biopsied no sooner than 2 weeks prior to treatment.
4. Patients who may have high burden of disease (i.e., large lesions), who are non-surgical candidates or who refuse surgery.
5. Non-surgical candidates, who may be able to undergo resection of selected single, individual lesion, but may not tolerate extensive surgery, may have many co morbidities, may be prone to complications.
6. Patients in whom surgery or radiation therapy may be impractical.
7. Primary lesions may be acceptable for enrollment.
8. Within normal limit hematopoietic capacity, hepatic and renal function. Values outside those limits may be allowed at the discretion of the PI, if they are determined as not clinically significant.
9. Evidence of a personally signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.
10. Ability to understand and the willingness to sign a written informed consent document in English.

Exclusion Criteria

Patients will be excluded from the study based on the following criteria:

1. Sexually active women of childbearing (WOCBP)* who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for 20 months after the final dose of treatment. Highly effective contraceptive measures include:

   1. Stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation
   2. Intrauterine device (IUD); intrauterine hormone-releasing system
   3. Bilateral tubal ligation;
   4. Vasectomized partner (provided that the vasectomized partner is the sole sexual partner of the WOCBP study subject);
   5. and/or sexual abstinence.

      * Childbearing potential refers to a female who has reached menarche, has not had a surgical sterilization procedure (such as a hysterectomy or bilateral oophorectomy), and is not postmenopausal. Menopause is defined as 12 consecutive months of amenorrhea without other biological causes. Furthermore, for females under 55 years old, a serum follicle-stimulating hormone level greater than 40 mIU/mL must be documented to confirm menopause.
2. Sexually active males who are unwilling to use a condom with female partners of childbearing potential, during the study, and for at least 8 months after the last dose of treatment.
3. Subjects who plan on donating blood or blood products during the study and for at least 20 months after the last dose of treatment. Male subjects must agree not to donate sperm during the study and for at least 8 months after the last dose of treatment.
4. Target lesions of basal cell carcinomas of aggressive subtypes (infiltrative, morpheaform, micronodular).
5. Any BCC that may require Mohs surgery for definitive control as a target lesion.
6. Subjects with porphyria's or known hypersensitivity to porphyrins.
7. Subjects with known photosensitivity diseases.
8. Subjects previously treated with a systemic photosensitizer within 4 months of screening date.
9. Subjects who desire to get pregnant a female of childbearing potential within the next 1.5 years.
10. Uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Life expectancy less than one year.
12. Inability or unwillingness to swallow capsules.
13. Have a history of alcohol of substance abuse, unless in full remission for greater than 6 months prior to the screening visit (Day 0) when the consent form is signed.
14. Having used any of the following treatment within 6 months before the baseline visit:

    * hedgehog pathway inhibitor, biologics, or chemotherapy
    * topical chemotherapy agents including Imiquimod, fluorouracil,) to the selected treatment lesion sites within 3 weeks.
15. Currently undergoing treatment with photodynamic therapy within 3 weeks before baseline visit.
16. Subjects who have received any type of solid organ transplant.
17. Subjects taking immunosuppressive medications at the screening visit that interact with Sonidegib at the screening visit unless approved by the investigator..
18. Participation in other study using an investigational or experimental therapy or procedure within 4 weeks or 5 half-lives (whichever is longer) before the screening visit and/or during study participation. Subjects cannot participate in studies of other investigational or experimental therapies or procedures at any time during their participation in this study.
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
20. Subjects unable or unwilling to comply with the study visit schedule and requirements of the study.
21. Subjects unable to speak and read the English language.
22. A subject who, in the opinion of the sponsor-investigator will be uncooperative or unable to comply with study procedures.
23. A subject who, in the opinion of the sponsor-investigator will be uncooperative or unable to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome | From enrollment to day 180
  Primary efficacy outcome measure: the overall response rate (ORR) to the combination therapy in patients, which is the proportion of evaluable study subjects who has complete response (CR) or partial response (PR) to the study treatment as defined in the protocol.
Review of AEs likely related to study drug | From enrollment to day 180
  Primary safety outcome measure: the proportion of evaluable study participants who had a grade 3 or higher adverse event (AE) or any serious adverse event (SAE) that determined to be at least possibly or probably related to study treatment, or any AE which is at least possibly or probably related to study treatment that causes permanent study discontinuation. The efficacy outcome measure: the overall response rate (ORR) to the combination therapy in patients, which is the proportion of evaluable study subjects who has complete response (CR) or partial response (PR) to the study treatment.

SECONDARY OUTCOMES:
Review of disease progression | From enrollment to day 180
  The secondary efficacy outcome measures: the proportion of evaluable subjects with progressive disease (PD), and the proportion of evaluable subjects with stable disease (SD). The proportion of evaluable study subjects who have complete histological clearance (CHC). The secondary safety outcome measures: the proportion of evaluable subjects who have AE of any specific grade or any specific type, or any SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Zeitouni, MD, Principal Investigator — Medical Dermatology Specialists
Locations (1):
- Medical Dermatology Specialists, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Contractual obligations with SunPharma

REFERENCES:
- [Background] Itkin A, Gilchrest BA. delta-Aminolevulinic acid and blue light photodynamic therapy for treatment of multiple basal cell carcinomas in two patients with nevoid basal cell carcinoma syndrome. Dermatol Surg. 2004 Jul;30(7):1054-61. doi: 10.1111/j.1524-4725.2004.30317.x. PMID 15209801
- [Background] Maytin EV, Kaw U, Ilyas M, Mack JA, Hu B. Blue light versus red light for photodynamic therapy of basal cell carcinoma in patients with Gorlin syndrome: A bilaterally controlled comparison study. Photodiagnosis Photodyn Ther. 2018 Jun;22:7-13. doi: 10.1016/j.pdpdt.2018.02.009. Epub 2018 Feb 19. PMID 29471147
- [Background] Lanoue J, Goldenberg G. Basal Cell Carcinoma: A Comprehensive Review of Existing and Emerging Nonsurgical Therapies. J Clin Aesthet Dermatol. 2016 May;9(5):26-36. Epub 2016 May 1. PMID 27386043
- [Background] Epstein EH. Basal cell carcinomas: attack of the hedgehog. Nat Rev Cancer. 2008 Oct;8(10):743-54. doi: 10.1038/nrc2503. PMID 18813320